CLINICAL TRIAL: NCT04633967
Title: Observational Study of a Novel Peri Infusion Regimen on the Infusion Associated Reactions With Alemtuzumab Infusion in Patients With Multiple Sclerosis in a Canadian Clinical Setting.
Status: Completed | Type: Observational
Sponsor: Maritime Neurology (Network)
Responsible Party: Sponsor
Other Study IDs: KesoKeso21
Record Dates: First submitted 2020-10-26; First posted 2020-11-18 (Actual); Last update posted 2024-03-13 (Actual); Status verified 2021-10

CONDITIONS: Frequency of Infusion Reactions in Novel Versus Standard Protocol in Multiple Sclerosis
MeSH Terms: interventions — Alemtuzumab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Drug: Alemtuzumab Injection — This observational study is collecting clinical data focusing on infusion associated reactions and changes in vital signs in MS patients Novel Infusion protocol: The protocol consisted of the following Pre-infusion Protocol
  Premedication with an H1 and H2 blockade (ranitidine or similar, loratadine or similar) for 7 days prior to the infusion.
  Premedication with 50 mg of prednisone orally for 5 days before the infusion.
  During Infusion Protocol During infusions methylprednisolone is administered in a dosage of 500 mg on every day of the infusion.
  Post Infusion Medication
  Post-medication with an H1 and H2 blockade (ranitidine or similar, loratadine or similar) for 7 days after the infusion.
  Post-medication with 50 mg of prednisone orally for 5 days after the infusion.
  Medications to be used PRN throughout the peri-infusion protocol Benadryl, acetaminophen or other analgesics were allowed

SUMMARY:
To evaluate a Novel infusion protocol in MS patients treated with Alemtuzumab

DETAILED DESCRIPTION:
This observational study will evaluate and anaylse primary data investigating the effects of a novel peri-infusion regimen in MS patients in a Candian clinical setting infused with Alemtuzumab.

This observational study has been developed by a Canadian neurologist with the intent to treat MS patients receiving Alemtuzumab in order to mitigate infusion associated reactions (safety) by utilizing an alternative peri-infusion protocol which is a deviation from the recommendation in the Canadian Product Monograph.

All the patients' recruited for this observational study were informed and consented for this novel peri-infusion regimen and were clinically followed by the neurologist for the two Alemtuzumab infusion cycles and for any subsequent Alemtuzumab infusions for potential mitigation of infusion associated reactions associated with Alemtuzumab.

ELIGIBILITY:
Inclusion Criteria: Patient s treated with Alemtuzumab as per canadian label -

Exclusion Criteria: Contraindication to Alemtuzumab

-

Ages: 18 Years to 65 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Adult patients with MS qualifying for Alemtuzumab therapy
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2016-05-15 (Actual); Primary Completion 2020-12-30 (Actual); Study Completion 2021-02-28 (Actual)

PRIMARY OUTCOMES:
Number and type of adverse events in Novel versus standard infusion protocol | 2016-2020
  This will include Changes In T,BP, R , during infusion, Need for extended observation, additional medication required or Neurological complications within 7 days of infusion , including headache, worsening of MS as measured by EDSS and peri-infusion infections.

CONTACTS AND LOCATIONS:
Locations (1):
- Maritime Neurology, Halifax, Nova Scotia, Canada

IPD SHARING:
Plan to Share IPD: No